CLINICAL TRIAL: NCT04043156
Title: RAdiotherapy for Metastatic Spinal Cord Compression with Increased Radiation DosES
Acronym: RAMSES-01
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 52 of 65 planned patients were recruited. Since during the study, survival was worse than expected, a new survival score was developed, which was more precise than the tool used for the RAMSES-01 trial. As a consequence, the trial was terminated.
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Prof Dirk Rades, Chair of the Department of Radiation Oncology, University of Luebeck, University Hopsital Schleswig Holstein Campus Lübeck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAMSES-01
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Compression Due to Metastasis to Spine
Keywords: spinal cord compression, radiotherapy
MeSH Terms: conditions — Spinal Cord Compression

STUDY DESIGN:
Intervention Model Description: Single arm study compared with a historical cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High-precision RT (Experimental): Study Arm: 18 x 2.33 Gy of high-precision RT in 3.5 weeks.
  Interventions: Radiation: High-precision RT

INTERVENTIONS:
Radiation: High-precision RT — 18 x 2.33 Gy of high-precision RT in 3.5 weeks

SUMMARY:
This clinical study aims to investigate whether high-precision radiotherapy, as supposed, leads to a better control of the irradiated spinal cord metastases when compared to conventional radiotherapy. This means that a progression or recurrence of motor deficits (weakness) of the legs following radiotherapy can be avoided more effectively. Furthermore, the high-precision radiotherapy will be compared to the conventional radiotherapy with respect to pain relief, motor function/ability to walk, quality of life, side effects and survival.

DETAILED DESCRIPTION:
The aim of this single-arm study is to show that high-precision radiotherapy (RT) with 18x2.33 Gy in 3.5 weeks results in significantly better local progression free survival (LPFS) of metastatic spinal cord compression (MSCC) when compared to conventional RT with 10x3 Gy in 2 weeks. If such superiority could be shown, 18x2.33 Gy could be recommended, at least for those patients with favourable survival prognoses, since an in-field recurrence of MSCC in the irradiated part of the spine is generally very difficult to treat.

For this investigation the newly prospectively collected data will be compared with a historical cohort collected up to the time of data analysis.

The recruitment of all 65 patients (62 patients + 5% for potential drop-outs) is planned to be completed within 21 months. The follow-up period will be 12 months. This equals a total running time for the study of 33 months.

In accordance with a previous study assessing local control of MSCC, the following patient characteristics will be recorded to allow adequate comparison with the historical control group:

* Age
* Gender
* Type of primary tumor (breast cancer vs. prostate cancer vs. myeloma/ lymphoma vs. lung cancer vs. other tumors)
* Interval from tumor diagnosis to MSCC (≤15 months vs. >15 months)
* Number of involved vertebrae (1-2 vs. ≥3)
* Other bone metastases at the time of RT (no vs. yes)
* Visceral metastases at the time of RT (no vs. yes)
* Time developing motor deficits prior to RT (1-7 days vs. 8-14 days vs. >14 days)
* Ambulatory status prior to RT (no vs. yes)
* Eastern Cooperative Oncology Group (ECOG) performance score (0-2 vs- 3-4)
* Indication for decompressive surgery of affected spinal areas

The patients of this study who received high-precision RT with 18x2.33 Gy for MSCC will be compared to a historical control group of patients with a favorable survival prognosis who were treated with 10x3 Gy of conventional RT. The historical control group will include data from 235 patients qualifying for the comparison with the prospectively collected data.

Data for the historical control group will be collected from an already existing anonymized database with previous study data documented in the European Union.

To be eligible for control group, patients fulfilling the same inclusion criteria and exclusion criteria as defined in the prospective study are considered. Furthermore, to be consistent with efficacy analysis of the study, patients of the historical control group must have received at least 80% of the planned RT dose.

Propensity score techniques will be applied to reduce confounding due to differences between the historical control group and the prospective trial data.

ELIGIBILITY:
Inclusion Criteria:

1. Motor deficits of the lower extremities resulting from MSCC, which have persisted for no longer than 30 days
2. Confirmation of diagnosis by MR-imaging (computed tomography [CT] allowed)
3. Age 18 years or older
4. Written informed consent
5. Favorable survival prognosis (defined as 36-45 points on the survival score)
6. Capacity of the patient to contract

Exclusion Criteria:

1. Previous RT or surgery of the spinal areas affected by MSCC
2. Symptomatic brain tumor or symptomatic brain metastases
3. Metastases of the cervical spine only
4. Other severe neurological disorders
5. Pregnancy, Lactation
6. Clear indication for spinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Local progression-free survival at 12 months following RT. | For each patient 12 months after the end of RT.
  LPFS time will be calculated from the last day of the RT. The evaluation will be performed in those patients, who are available for assessement of the Primary endpoint and have received at least 80% of the planned RT dose.

SECONDARY OUTCOMES:
Change in motor function/ability to walk | Assessment directly and at 1, 3, 6, 9 and 12 months after RT.
  Change in motor function is defined as improvement or deterioration by at least one point. 0=normal strength; 1=ambulatory without aid; 2 ambulatory with aid; 3=not ambulatory;4=complete paraplegia. Motor function will additionally be evaluated using additionally the American Spinal Injury Association (ASIA) classification resulting in total points of 0 to 14.
Change in quality of life | Evaluation directly and at 1, 3, 6, 9 and 12 months after RT
  Quality of life (QoL) will be assessed using the distress thermometer. Patients can rate their impairment in QoL between 0 and 10 (no to maximum impairment). The data will be compared to the data documented prior to RT
Change in vertebral pain | Evaluation directly and at 1, 3, 6, 9 and 12 months after RT
  Vertebral pain will be evaluated with a numeric rating scale (self-assessment by patients ) from 0=no pain to 10=worst pain. Improvement by 2 points is rated partial response, 0 points complete response. The data will be compared to the data documented prior to RT. The intake of analgesics will be included.
Overall survival | Evaluation directly and at 1, 3, 6, 9 and 12 months after RT
  Will be calculated from the last day of RT up to 12 months following RT.
Local progression-free survival | Additional evaluation directly and 1, 3, 6 and 9 months after RT
  LPFS time will be calculated from the last day of the RT.
Occurence of toxicity | Evaluation during RT and directly, 1, 3, 6, 9 and 12 months after RT
  Toxicity will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) 4.3. If radiation myelopathy is suspected, spinal Magnetic Resonance (MR)-Imaging will be performed. The data will be compared to the data documented prior to RT.
Change in sensory function | Evaluation during RT and directly, 1, 3, 6, 9 and 12 months after RT
  Sensory function will be evaluated using the following scale, modified in accordance to the ASIA classification, 0=absent, 1=impaired, 2=normal, 9=cannot be assessed.
Chance in sphincter dysfunction | Evaluation during RT and directly, 1, 3, 6, 9 and 12 months after RT
  Sphincter dysfunction will be evaluated as yes versus no.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, Prof. Dr., Principal Investigator — Dep. of Radiation Oncology, Univ. of Lübeck and Univ. Medical Center S-H
Locations (1):
- Department of Radiation Oncology, University of Lübeck and University Medical Center Schleswig-Holstein, Ratzeburger Allee 160, 23562 Lübeck, Germany, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rades D, Hansen O, Jensen LH, Dziggel L, Staackmann C, Doemer C, Cacicedo J, Conde-Moreno AJ, Segedin B, Ciervide-Jurio R, Rubio-Rodriguez C, Perez-Romasanta LA, Alvarez-Gracia A, Dennis K, Ferrer-Albiach C, Navarro-Martin A, Lopez-Campos F, Jankarashvili N, Janssen S, Olbrich D, Hollander NH. Radiotherapy for metastatic spinal cord compression with increased radiation doses (RAMSES-01): a prospective multicenter study. BMC Cancer. 2019 Nov 29;19(1):1163. doi: 10.1186/s12885-019-6390-x. PMID 31783816